CLINICAL TRIAL: NCT01521910
Title: Effect of Dietary Protein Restriction on Prognosis in Patients With Diabetic Nephropathy
Acronym: LPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Peter Rossing, Chief physician and Director of Research, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Low Protein Diet
Record Dates: First submitted 2012-01-13; First posted 2012-01-31 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Type 1 Diabetes Mellitus With Diabetic Nephropathy
Keywords: survival; protein restriction; diabetic nephropathy; type 1 diabetes; GFR; ESRD; progressive renal disease
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 1; Kidney Failure, Chronic | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low protein diet (Experimental)
  Interventions: Dietary Supplement: low protein diet
- Normal protein diet (Active Comparator)
  Interventions: Dietary Supplement: normal protein diet

INTERVENTIONS:
Dietary Supplement: low protein diet — An iso-caloric low protein diet of 0.6 g/kg/day was prescribed during the whole study duration.
  The same dietician gave nutritional advices at least every three months during the whole study period. Patients were also seen by the same doctor during each visit for the whole study period.
  Supplementation of Calcium of 500mg/day.
  Urine albumin losses >= 2 g/day wre replaced by increasing dietary protein on a gram-for-gram basis, only if the patient was compliant with the prescribed low-protein diet.
  Arms: Low protein diet
Dietary Supplement: normal protein diet — The patients pre-study diet during the whole study period
  Patients were also seen by the same doctor during each visit for the whole study period.
  Arms: Normal protein diet

SUMMARY:
The purpose of the investigators study was to determine the effect of dietary protein restriction on survival and progression to end stage renal disease (ESRD) in diabetic nephropathy.

DETAILED DESCRIPTION:
The study was a prospective, randomized, unmasked, controlled trial carried out at the Steno Diabetes Center. With concealed randomization the patients were (in blocks of two according to the level of GFR) assigned to receive either a usual-protein diet or a low-protein diet.

After randomization an iso-caloric low-protein diet of 0.6 g/kg/day was prescribed to patients in the low-protein diet group. The usual-pro tein diet consisted of the patients' pre-study diet.

The planned duration of follow-up was four years, scheduled visits every three-months. All patients gave complete history of medication, underwent examination of weight, urinary albumin-, sodium- and urea excretion, serum albumin, serum urea, hemoglobin, hemoglobin A1c, blood pressure, serum total-cholesterol, high-density lipoprotein (HDL) cholesterol.

GFR, serum triglycerides,calcium and phosphorous, anthropometric measurements, nutritional status and smoking habits were evaluated every six months.

Dietary protein intake was estimated on the basis of three consecutive 24-hour urine samples completed before each visit, using urinary excretion of urea nitrogen.

GFR was measured by plasma clearance of 51Cr-EDTA over a 4 hour period and standardized for 1.73m2 body surface area using the same surface for each patient during the study.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 1
* duration at least 10 years
* onset before age of 35,
* presence of diabetic retinopathy
* albuminuria>=300mg/24 h in at least 2/3 sterile urine samples
* no clinical or laboratory evidence of other kidney or urinary tract disease
* GFR above 20mL/min/1.73M2
* pre-study decline in GFR>= 2 mL/min/year

Exclusion Criteria:

* pregnancy
* history of congestive heart failure or myocardial infarction or coronary bypass surgery within the last three months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 1995-04; Primary Completion 2000-06 (Actual); Study Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of ESRD requiring dialysis or transplantation, and death | 4 years
  Cause of death was obtained from death certificate by an independent observer. Before the development of uremic symptoms, patients were referred to the department of nephrology at the University Hospital of Herlev or Rigshospitalet, when GFR deteriorated below 10 to 20 ML/min/1.73m2, where accepted criteria for initiation of dialysis and transplantation were applied on patients from both diet groups. Patients continued their scheduled visits and treatment in the study until the end of the four-year follow up.
  This was assesed every 3 months until the end of the 4 year follow up period.
Rate of decline of GFR | 4 years
  rate of decline was measured if the patient had a minimum of one year of follow up and a minimum of 3 GFR measures during the study. All measures of GFR during the study period (including baseline) were used to calculate the rate of decline(the slopes) of GFR. GFR was measured every 6 months during the 4 years of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik P Hansen, MD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Gentofte, Denmark